CLINICAL TRIAL: NCT01744340
Title: A Dose Finding Study of Eribulin Mesylate and Cetuximab For Patients With Advanced Head and Neck and Colon Cancer With an Expansion Cohort For Head and Neck Cancer: A Brown University Oncology Research Group Study
Brief Title: A Dose Finding Study of Eribulin Mesylate and Cetuximab For Patients With Advanced Head and Neck and Colon Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: howard safran (Other)
Collaborators: Fatima Memorial Hospital (Other); Montefiore Medical Center (Other); Rhode Island Hospital (Other); The Miriam Hospital (Other)
Responsible Party: Sponsor-Investigator, howard safran, Prinicipal Investigator, Brown University
Organization: Brown University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG 254
Record Dates: First submitted 2012-02-23; First posted 2012-12-06 (Estimated); Results first posted 2016-02-10 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Head and Neck Cancer; Colon Cancer
Keywords: Head and Neck; Colon
MeSH Terms: conditions — Head and Neck Neoplasms; Colonic Neoplasms | interventions — TNFAIP8 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- head and neck (Experimental): Cetuximab, 400 mg/m2 cycle 1 week 1, then 250 mg/m2/weekly there after Eribulin Mesylate 1.4mg/m2
  Interventions: Drug: Head and neck
- Colon- closed as of May 2014 (Experimental): Eribulin Mesylate:
  1.4 mg/m2 IV infusion days 1 and 8 of 21 day cycle
  Interventions: Drug: Colon- Closed as of May 2014

INTERVENTIONS:
Drug: Head and neck — Eribulin mesylate is administered by IV infusion over 2-5 minutes on day 1 and 8 of a 21 day cycle 1.4mg/m2 and Cetuximab 400 mg/m2 cycle 1 week 1, then 250 mg/m2/weekly thereafter
  Dose Level 1: 0.7 mg/m2 IV infusion days 1 and 8 of 21 day cycle Dose Level 2: 1.0 mg/m2 IV infusion days 1 and 8 of 21 day cycle Dose Level 3: 1.4 mg/m2 IV infusion days 1 and 8 of 21 day cycle
  Arms: head and neck
Drug: Colon- Closed as of May 2014 — Eribulin Mesylate:
  1.4 mg/m2 IV infusion days 1 and 8 of 21 day cycle
  Arms: Colon- closed as of May 2014

SUMMARY:
The purpose of this study is to determine if the full dose of eribulin mesylate can be safely given with the full dose of cetuximab. The activity of the combination of eribulin mesylate and cetuximab on recurrent head and neck cancer and colon cancer will also be assessed.

DETAILED DESCRIPTION:
To determine if eribulin mesylate, up to a maximum dose of 1.4 mg/m2 day 1 and 8 of a 21 day cycle, can be safely combined with full dose cetuximab for patients with advanced head and neck cancer and colon cancer

ELIGIBILITY:
Inclusion Criteria

* Histologically or cytologically confirmed advanced squamous cell cancer of the head and neck with progression after at least one prior therapy. (Chemoradiation is considered one line of therapy). Patients with unknown Head and Neck primaries are also eligible
* In the dose escalation cohorts, patients with advanced colon adenocarcinoma with wild-type kras who have previously received at least two lines of therapy for advanced disease are eligible- No longer applicable post February 2013 as all patients have been enrolled to the dose escalation phase
* In the expansion phase for patients with advanced colorectal cancer, only patients with mutated kras who have previously received at least two lines of therapy for metastatic disease will be eligible. Pathology report from diagnosis and report documenting KRAS status to be sent to BrUOG. No longer applicable as this phase of the study has been closed as of 5/6/2014 secondary to the lack of efficacy and activity of the single agent.
* Life expectancy of at least 3 months
* Patients must be aged 18 years or older
* Patients with measurable tumors according to RECIST .
* Patients must have an Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
* No severe concurrent illness that would interfere with protocol therapy.
* Patients must have adequate renal function as evidenced by ≤1.5 mg/dL or creatinine clearance > 40 mL/minute (min).
* Patients must have adequate bone marrow function as evidenced by absolute neutrophil count (ANC) > 1.5 x 109/L and platelet count > 100 x 109/L.
* Patients must have adequate hepatic function as evidenced by bilirubin ≤ 1.5 times the upper limit of normal (ULN) and alanine aminotransferase (ALT), and aspartate aminotransferase (AST) ≤ 3 x ULN (in the case of liver metastases ALT and AST ≤ 5 x ULN).
* Resolution of all chemotherapy or radiation-related toxicities to Grade 1 severity or below, except for alopecia.
* Patients must be willing and able to comply with the study protocol for the duration of the study.
* Patients must give written informed consent prior to any study-specific screening procedures with the understanding that the patient may withdraw consent at any time without prejudice.
* No other active invasive malignancy unless disease free for at least 2 years.

Exclusion Criteria

* For Head and Neck patients, no progression while receiving an EGFR inhibitor or within 6 months of stopping treatment with an EGFR inhibitor.
* Patients who received chemotherapy or investigational therapy within 3 weeks before treatment initiation. Radiation must be completed within 2 weeks before treatment initiation.
* Patients with a hypersensitivity to halichondrin B and/or halichondrin B chemical derivative.
* Patients who participated in a prior eribulin mesylate clinical trial, whether or not they received eribulin mesylate.
* Patients with other significant disease or disorders that, in the investigator's opinion, would exclude the patient from the study.
* Women who are pregnant or breast-feeding; women of childbearing potential with either a positive pregnancy test at screening or no pregnancy test; women of childbearing potential unless (1) surgically sterile or (2) using adequate measures of contraception in the opinion of the Investigator. Peri-menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential.
* Patients with brain or subdural metastases are not eligible, unless they have completed local therapy and have discontinued the use of corticosteroids for this indication for at least 4 weeks before starting treatment in this study. Any signs (e.g., radiologic) and/or symptoms of brain metastases must be stable for at least 4 weeks.
* Grade 2 or worse neuropathy.
* Significant cardiovascular impairment (history of congestive heart failure > NYHA G II, unstable angina or myocardial infarction within the past six months, or serious cardiac arrhythmia.
* QTc > 500 msec

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-05; Primary Completion 2015-03 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Safran, MD, Principal Investigator — Brown University
Locations (4):
- United States (4):
  - Montefiore, The Bronx, New York
  - Memorial Hospital, Pawtucket, Rhode Island
  - Rhode Island Hospital, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island

RESULTS

PARTICIPANT FLOW:
Groups:
- Head and Neck: Cetuximab, 400 mg/m2 cycle 1 week 1, then 250 mg/m2/weekly there after Eribulin Mesylate 1.4mg/m2
  Head and neck: Eribulin mesylate is administered by IV infusion over 2-5 minutes on day 1 and 8 of a 21 day cycle 1.4mg/m2 and Cetuximab 400 mg/m2 cycle 1 week 1, then 250 mg/m2/weekly thereafter
  Dose Level 1: 0.7 mg/m2 IV infusion days 1 and 8 of 21 day cycle Dose Level 2: 1.0 mg/m2 IV infusion days 1 and 8 of 21 day cycle Dose Level 3: 1.4 mg/m2 IV infusion days 1 and 8 of 21 day cycle
- Colon- Closed as of May 2014: Eribulin Mesylate:
  1.4 mg/m2 IV infusion days 1 and 8 of 21 day cycle
  Colon- Closed as of May 2014: Eribulin Mesylate:
  1.4 mg/m2 IV infusion days 1 and 8 of 21 day cycle
Period: Overall Study
Arm/Group | Head and Neck | Colon- Closed as of May 2014
Started | 8 | 15
Completed | 8 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Head and Neck | Colon- Closed as of May 2014 | Total
Number analyzed (Participants) | 8 | 15 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 9 | 14
  >=65 years | 3 | 6 | 9
Age, Continuous [Mean (Full Range); unit: years] | 58.5 [45 to 70] | 71 [41 to 86] | 60.6 [41 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 8 | 8
  Male | 8 | 7 | 15
Region of Enrollment [Number; unit: participants]
  United States | 8 | 15 | 23

OUTCOME MEASURES:

1. Primary Outcome: If Eribulin Mesylate, up to a Maximum Dose of 1.4 mg/m2 Day 1 and 8 of a 21 Day Cycle, Can be Safely Combined With Full Dose Cetuximab for Patients With Advanced Head and Neck Cancer and Colon Cancer.
Description: A DLT was defined as:
  * Grade 4 neutropenia (ANC < 500/mm3) for > 7 days
  * ANC <1000/mm3 with fever or infection
  * Platelets <25,000/mm3
  * Platelets <50,000/mm3 requiring transfusion
  * Grade 3 or grade 4 treatment related non-hematologic toxicities excluding alopecia. Grade 3 nausea, vomiting or diarrhea will only be considered a dose limiting toxicity if it occurs despite maximal medical support. Grade 3 or grade 4 hypomagnesemia will not be considered a dose limiting toxicity since it is an expected side effect of cetuximab and can be corrected. Other grade 3 or grade 4 electrolyte abnormalities will not be considered dose limiting toxicities if the electrolyte disorder can be corrected to grade 2 or less within 72 hours.
  * EGFR dermatologic toxicity should be graded according to the toxicity scale for EGFR associated reactions. The first episode of grade 3 or grade 4 rash will not be considered a DLT.
  * If any patient receives < 70% of the planned dose of eribulin mesylat
Time Frame: From Day 1 of Drug through end of cycle 2 equals (approximately) 42 days
Population: Outcome measure that address the dose of 1.4 mg/m2,6 patients were treated (1 head and neck 5 colon). 12 patients were enrolled in the course of the MTD dose finding,10 colon and 2 head and neck. All other results sections are inclusive of all patients(dose finding +expansion cohort).
Measure: Number; unit: participants
Arm/Group | Head and Neck | Colon- Closed as of May 2014
Number analyzed (Participants) | 1 | 5
participants | 0 | 0

2. Secondary Outcome: Response Rate (Whether Patient's Disease is Progressing or Being Controlled) of Patients With Head and Neck Cancer Treated With Eribulin Mesylate and Cetuximab.
Description: This shows patients able to achieve Stable disease or better as their best response during course of study participation. Response will be evaluated by Revised Response Evaluation Criteria in Solid Tumors (RECIST) Guideline v1.1 RECIST Guideline version 1.1 Response Criteria Complete Response:Disappearance of all target lesions; Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial Response: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters Progressive Disease:At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
  Stable Disease:Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study
Time Frame: From beginning of treatment to progression of disease, for an expected average of 1 year
Measure: Number; unit: participants
Arm/Group | Head and Neck | Colon- Closed as of May 2014
Number analyzed (Participants) | 8 | 15
participants | 6 | 2

ADVERSE EVENTS:
Time Frame: Adverse events were collected pre-study, within 72 hours of day 1 if each cycle, at day 8 of each cycle, at end of treatment visit and 30 days post last dose of drug.
Arm/Group | Head and Neck | Colon- Closed as of May 2014
Serious Adverse Events (participants affected / at risk) | 5/8 | 1/15
Other Adverse Events (participants affected / at risk) | 8/8 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Head and Neck (N=8) | Colon- Closed as of May 2014 (N=15)
S b(4), pleural effusion(4), Dyspnea(4), asp(4), lung inf (4), resp acidosis(4) (Investigations) | 1 (1) | 0 (0) — Shortness of breath (4), left pleural effusion (4) , Dyspnea (4), aspiration (4), lung infection (4), resp acidosis(4)
Acute respiratory failure (5) (Investigations) | 1 (1) | 0 (0)
Dyspnea(2), K(3) , MG(2) , ANC(3), Nausea(2), Vomitting(2) (Investigations) | 1 (1) | 0 (0)
Edema(3), dysphyagia(3), hemolytic Anemia(3), PLT(4), calcium(1),WBC(1) , lymph(3) (Investigations) | 1 (1) | 0 (0)
Hemorragic shock(5), HGB/Anemia(3), Chloride(1) , CO2(1) , AST(2), ALT(2) , PT(1) (Investigations) | 1 (1) | 0 (0)
COPDdyspnea(2),neutr(3),sepsis(4),anemia(2),Leuk(3),Lymph (3), Hypergly(2),Hypoca(2), Hypokal(1) (Investigations) | 1 (1) | 0 (0) — COPD exasp dyspnea (2), neutropenia(3), sepsis(4), anemia (2), Leukopenia(3),Lymphocyte decrease(3), Hyperglycemia(2),Hypocalemia(2), Hypokalemia(1)
Dyspnea(1), Sepsis(4), Anemia(2), Lymphocyte decrease (3), Hypocalcemia(2) (Investigations) | 1 (1) | 0 (0)
Feb neut(3), neut(4),anemia(3), leuk(3),hypona(3), lymph(3) , CR(1), Ca(2), K(1), Gluc(1), MG(2) (Investigations) | 1 (1) | 0 (0) — Febrile neutropenia(3), neutropenia (4),anemia(3), leukopenia(3),hyponatremia(3) , lymphocyte count(3) , CR(1), Calcium(2), K (1), Gluc(1), MG(2)
Feb Neut(res).Neut(0),An(1),Leuk(0),Hypona(1),Lymph(1),CR(0),Ca(1),K(0),Gluc(0),MG(1),URI(2)O Muc(3) (Investigations) | 1 (1) | 0 (0) — Febrile Neutropenia (resolved). Neutropenia(0), Anemia(1), Leukopenia(0), Hyponatremia(1), Lymphocyte count(1), CR(0), Calcium(1), K(0), Gluc(0), MG(1),URI(2) , Oral Mucositis(3)
Respiratory Infection (5) (Investigations) | 1 (1) | 0 (0)
Dyspnea(2), Febrile Neutropenia(3) (Investigations) | 1 (1) | 0 (0)
Dyspnea(2), Productive cough(2), Wheezing(3) (Investigations) | 1 (1) | 0 (0)
Dys(1),PrCo(0),Whez(0),Resp(4),An(3),HGB(3),Leuk(1),Lymph(3),ALB(2),CA(2),K(3),MG(2),PHOS(4),GLU(2) (Investigations) | 1 (1) | 0 (0) — Dyspnea (1), Productive Cough (0), Wheezing (0), Respiratory failure (4), Anorexia (3), HGB(3), Leukopenia(1), Lymph(3), HypoALB(2), CA(2), K(3), MG(2), PHOS(4), GLU(2)
Na(3), confusion(1), Fatigue(3), constipation(2), anorexia(3) (Investigations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Head and Neck (N=8) | Colon- Closed as of May 2014 (N=15)
Albumin (Investigations) | 7 (7) | 7 (7)
Allergic Rhinitis (Investigations) | 1 (1) | 0 (0)
ALK (Investigations) | 0 (0) | 2 (2)
ALT (Investigations) | 2 (2) | 5 (5)
Alopecia (Investigations) | 2 (2) | 2 (2)
Absolute Neutrafil Count (Investigations) | 1 (1) | 6 (6)
anemia/HGB/Hemolytic anemia (Investigations) | 5 (5) | 7 (7)
Anorexia (Investigations) | 3 (3) | 2 (2)
Anxiety (Investigations) | 0 (0) | 1 (1)
AST (Investigations) | 2 (2) | 4 (4)
arterial blood gas (Investigations) | 1 (1) | 0 (0)
Bilirubin (Investigations) | 0 (0) | 2 (2)
blurry vision (Investigations) | 0 (0) | 1 (1)
bleed-urination (Investigations) | 1 (1) | 0 (0)
bloat/dyspepsia (Investigations) | 0 (0) | 2 (2)
Calcium (Investigations) | 2 (2) | 1 (1)
Chills (Investigations) | 2 (2) | 1 (1)
Constipation (Investigations) | 0 (0) | 3 (3)
Cough/Productive cough (Investigations) | 2 (2) | 0 (0)
Creatinine (Investigations) | 1 (1) | 1 (1)
CO2 (Investigations) | 1 (1) | 0 (0)
Chloride (Investigations) | 1 (1) | 0 (0)
Dehydration (Investigations) | 2 (2) | 1 (1)
Depression (Investigations) | 1 (1) | 1 (1)
Dizziness (Investigations) | 3 (3) | 1 (1)
Diarrhea (Investigations) | 2 (2) | 2 (2)
dry skin/pruritis/itching (Investigations) | 0 (0) | 3 (3)
Dysgeusia (Investigations) | 0 (0) | 1 (1)
Dysphagia (Investigations) | 1 (1) | 0 (0)
dry mouth (Investigations) | 2 (2) | 0 (0)
EGFR (Investigations) | 1 (1) | 0 (0)
erythema (periorbital, ear,facial flushing) (Investigations) | 1 (1) | 2 (2)
Fatigue (Investigations) | 7 (7) | 9 (9)
Fever (Investigations) | 1 (1) | 2 (2)
Glucose (Investigations) | 2 (2) | 0 (0)
H/A (Investigations) | 2 (2) | 4 (4)
hemoptysis (Investigations) | 1 (1) | 0 (0)
hypersensitivity rxn (Investigations) | 0 (0) | 2 (2)
Hypotension (Investigations) | 2 (2) | 1 (1)
infection (Investigations) | 1 (1) | 4 (4) — (eye, lung, mucosal, skin, parasitic, cellulitis g-tube, sepsis, Upper respiratory, thrush )
Irritability (Investigations) | 0 (0) | 1 (1)
Insomnia (Investigations) | 1 (1) | 1 (1)
Potassium (Investigations) | 5 (5) | 7 (7)
Lymphopenia/Lymphocytes (Investigations) | 3 (3) | 4 (4)
m/a (myalgia), weakness (Investigations) | 4 (4) | 0 (0)
Magnesium (Investigations) | 3 (3) | 1 (1)
muscle cramps (Investigations) | 1 (1) | 1 (1)
Mucositis, tongue and general (Investigations) | 4 (4) | 2 (2)
Sodium (Investigations) | 7 (7) | 3 (3)
nausea (Investigations) | 3 (3) | 4 (4)
neuropathy (Investigations) | 3 (3) | 3 (3)
sores mouth/lips (Investigations) | 0 (0) | 1 (1)
pain (general, abd,back,rib, chest, jaw, mouth,throat, hand, neck, head) (Investigations) | 5 (5) | 4 (4)
pericardial effusion (Investigations) | 1 (1) | 0 (0)
PT lab (Investigations) | 1 (1) | 0 (0)
Rash, acneform, pistula (Investigations) | 5 (5) | 7 (7)
rectal bleed/GI hemorrhage (Investigations) | 0 (0) | 2 (2)
Shortness Of Breath/dyspnea (Investigations) | 0 (0) | 1 (1)
thrombocytopenia (Investigations) | 0 (0) | 1 (1)
trismus (Investigations) | 1 (1) | 0 (0)
troponin (Investigations) | 1 (1) | 0 (0)
vomitting (Investigations) | 3 (3) | 2 (2)
watery eyes (Investigations) | 0 (0) | 1 (1)
White Blood Cells/leukopenia (Investigations) | 3 (3) | 9 (9)
wt loss (Investigations) | 5 (5) | 2 (2)
Phosphorus (Investigations) | 3 (3) | 0 (0)
sleep disorder (Investigations) | 1 (1) | 0 (0)
chest tightness (Investigations) | 1 (1) | 0 (0)
Hypoxemia (Investigations) | 1 (1) | 0 (0)
Delirium (Investigations) | 1 (1) | 0 (0)
Vision loss (Investigations) | 1 (1) | 0 (0)
DVT (Investigations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No